CLINICAL TRIAL: NCT06533566
Title: Effect of Erector Spinae Plane Block Versus Local Wound Infiltration on Postoperative Pain After Modified Radical Mastectomy
Brief Title: Erector Spinae Plane Block Versus Local Wound Infiltration After Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: pain after mastectomy
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain; Erector Spinae Plane Block; Local Infiltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Block (Active Comparator): Patients of this group will receive ultrasound guided erector spinae block with injection of (20 ml) of plain bupivacaine 0.25% (max dose 2mg/kg) injected beneath the erector spinae muscle sheath at the level of the fourth transvers process (T4).
  Interventions: Procedure: Erector spinae plane block
- Drain block (Active Comparator): Patients of this group will receive local wound infiltration (drain block) with injection of (20 ml) of plain bupivacaine 0.25% (max dose 2mg/kg) injected in each surgical drain (pectoral and axillary drains) thereafter, the drains would then clamped for 20 minutes and declamped later on.
  Interventions: Procedure: local wound infiltration

INTERVENTIONS:
Procedure: Erector spinae plane block — patients will be placed in the lateral decubitus position. The ESP block is usually performed at the level of fourth transvers process. The ultrasound probe should be placed in a cephalo-caudal orientation over the midline of the back at the desired level.Under aseptic conditions, the block needle will be inserted in plane at an angle of 30-40° in cranial-to-caudal direction until the tip contacted the T4 transverse process at erector spinae plane. After hydro-dissection with 2-3 mL of isotonic saline solution to confirm the correct needle tip position and after negative aspiration to prevent intra vascular injection or position, (20 ml) of plain bupivacaine 0.25% will be injected deep to the erector spinae muscle.
  Arms: Erector Spinae Block
Procedure: local wound infiltration — after the surgeon complete the surgery and insert the surgical drains (pectoral and axillary drains) we will inject 20ml of plain bupivacaine 0.25% in each surgical drain, the drains will be clamped for 20 minutes then declamped.
  Other Names: drain block
  Arms: Drain block

SUMMARY:
This randomized prospective double blinded study will aim to evaluate the postoperative analgesic effect of ultrasound guided Erector Spinae plane block and local wound infiltration (drain block) for patients scheduled for modified radical mastectomy surgery.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer worldwide and it represents 1 in 4 cancers diagnosed among women globally. Modified Radical Mastectomy (MRM) is a commonly performed surgery for breast cancer and is associated with moderate-to-severe postoperative pain. Poor postoperative pain management can lead to increased chances of the development of chronic pain. Therefore, adequate postoperative pain management after breast cancer surgery is essential. Regional block for pain management has many advantages in such patients including provision of adequate analgesia, reduced need for opioids, decreased postoperative nausea & vomiting and postoperative pulmonary complications. It also facilitates early ambulation. Thoracic Epidural (TE), paravertebral block (PVB), pectoral nerve I & pectoral nerve II blocks, serratus anterior plane block and erector spinae plan block have been used with good results. In particular, the erector spinae has proven to reduce pain severity and opioid consumption in this group of patients. Further, in meta-analysis, the ESP block was shown to effectively alleviate postoperative pain severity and reduce opioid consumption. In ESP block, local anesthetic is deposited deep to the erector spinae muscle which results in blocking of the ventral and dorsal rami of multiple spinal nerves. The LA diffuses into the paravertebral space and cephalo-caudally and blocks the pain by action on dorsal rami, ventral rami, and lateral cutaneous branches of intercostal nerves. Also, in many situations, a superior postoperative analgesia yet avoiding the detrimental effects of opioids, can be extracted from a simple technique of wound instillation of local anesthetics through surgical drain which provide a satisfactory long opioid free postoperative analgesic period.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-II
* scheduled for unilateral Modified radical mastectomy

Exclusion Criteria:

* Patient refusal.
* Patient with neurological deficit.
* Patient with bleeding disorders.
* Uncooperative patient.
* Infection at the block injection site.
* Patients with history of allergy to local anesthetics.
* Advanced hepatic, cardiac or renal failure.
* Chronic opioid consumption.
* Body mass index (BMI)≥ 30 kg m-2
* Chronic use of gabapentin or pregabalin

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 37 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | first postoperative day after modified radical mastectomy surgery
  total morphine amount which will be consumed in the first postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No